CLINICAL TRIAL: NCT04054973
Title: An Open-label Feasibility Trial of Adjunctive L-arginine and Tetrahydrobiopterin Combination in Patients With Treatment Resistant Schizophrenia
Brief Title: L-arginine Study for Persistent Symptoms of Schizophrenia
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was unable to be started due to unavailability of study medication.
Sponsor: University of Massachusetts, Worcester (Other)
Responsible Party: Principal Investigator, Xiaoduo Fan, Director, Psychotic Disorders Program, University of Massachusetts, Worcester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H00017202
Record Dates: First submitted 2019-08-02; First posted 2019-08-13 (Actual); Last update posted 2022-01-20 (Actual); Status verified 2022-01

CONDITIONS: Schizo Affective Disorder; Schizophrenia
Keywords: psychosis; Treatment resistant; L-arginine; MRS
MeSH Terms: conditions — Psychotic Disorders; Schizophrenia | interventions — Arginine; sapropterin

STUDY DESIGN:
Intervention Model Description: Open-label single arm pilot trial of L-arginine and Kuvan combination therapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- L-arginine and Kuvan (Experimental): Open-label single arm study, all participants will be in this group
  Interventions: Drug: L-arginine; Drug: Sapropterin Dihydrochloride

INTERVENTIONS:
Drug: L-arginine — 6000mg of L-arginine daily for 14 days
Drug: Sapropterin Dihydrochloride — 800mg of Kuvan daily for 14 days
  Other Names: Kuvan

SUMMARY:
The purpose of this research is to see if daily combination treatment of L-arginine and Kuvan changes brain chemistry in people experiencing schizophrenia as measured by MRS brain scans.

ELIGIBILITY:
Inclusion Criteria:

1. Males or Females aged 18-65 years inclusive.
2. English speaking.
3. Primary diagnosis of Schizophrenia established by a structured psychiatric evaluation (MINI) based on Diagnostic and Statistical Manual of Mental Disorders Fifth Edition (DSM-V) criteria.
4. Written informed consent in compliance with 21 CFR part 50 and in accordance with the International Conference on Harmonization (ICH) Good Clinical Practice (GCP) Guidelines.
5. A Positive and Negative Syndrome Scale (PANSS) (Kay et al 1987) total score ≥ 70 with a score of > 4 on two or more of the following PANSS items: delusions, conceptual disorganization, hallucinatory behavior, suspiciousness, and unusual thought content.
6. A score of ≥4 on the Clinical Global Impression-Severity (CGI-S) (Guy, 1976).
7. Must have ongoing antipsychotic treatment for at least 8 weeks, with a stable dose for at least 4 weeks. Antipsychotic medication will not be modified by the research team during the subject's enrollment or participation.
8. Subjects who have failed to achieve clinically-recognized symptom reduction to at least 1 marketed antipsychotic agent, given at a Physician Desk Reference (PDR)-defined therapeutic dose for ≥ 8 weeks during the past 12 months, will be eligible.
9. Women of childbearing potential must have a negative pregnancy test performed at screening visit prior to randomization. Women enrolled in this trial must use adequate birth control.
10. Understands and is able, willing, and (in the opinion of the investigator) likely to fully comply with the study procedures and restrictions.

Exclusion Criteria:

1. Subjects with a history of renal insufficiency, congestive heart failure, cardiac arrhythmias or history of myocardial infarction, liver cirrhosis, guanidinoacetate methyltransferase deficiency, herpes.
2. Subjects who are non-English speaking.
3. Subjects with any clinically significant abnormalities as determined by medical history, physical exam, clinical and lab evaluation suggestive of an underlying disease state that may, in the opinion of the investigator, confound the results of study, increase risk to the subject, or lead to difficulty complying with the protocol.
4. Subjects with the lab values defined as exclusionary safety values in Table 1.
5. On medications known to inhibit folate metabolism (e.g., methotrexate).
6. On medications known to affect NO-mediated vaso-relaxation (e.g., PDE-5 inhibitors such as sildenafil, vardenafil, or tadalafil).
7. Subjects on nitrates.
8. Subjects on levodopa.
9. Subjects on antihypertensive medications (such as ACE inhibitors, angiotensin receptor blockers, isoproterenol, potassium-sparing diuretics).
10. Subjects on antidiabetes medications.
11. Subjects on anticoagulant/antiplatelet medications.
12. Subjects with a current (within the last 3 months) DSM-V diagnosis of alcohol or substance use disorder (excluding nicotine and caffeine) as established by the clinical assessment (MINI) at the screening visit will be excluded.
13. Tested positive for the urine drug screen.
14. Subjects at imminent risk of suicide or injury to self or others, as per the opinion of the investigator, or history of significant suicide attempt within the last 6 months as per the Columbia Suicide Severity Rating Scale (C-SSRS).
15. Subjects that have taken an investigational drug or taken part in a clinical trial within 30 days prior to screening.
16. Known history of phenylketonuria (PKU).
17. Known hypersensitivity reactions (such as anaphylaxis and rash) to L-arginine and/or BH4.
18. Any other reason that, in the opinion of the investigator, would compromise patient safety or integrity of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-09-11 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Changes in brain chemistry as measured by 1H-MRS scans | 14 days
  To demonstrate that L-arginine and tetrahydrobiopterin (BH4) combination targets and alters brain chemistry in patients with TRS (target engagement). The investigators hypothesize that two-week treatment of L-arginine and Tetrahydrobiopterin (as Kuvan) will alter glutamate and GABA levels measured with proton magnetic resonance spectroscopy (1H-MRS).
Incidence of Treatment-Emergent Adverse Events as assessed by patient report | 14-days
  The study doctor in conjunction with the study coordinator will conduct a diagnostic interview with the subject at each visit to record the incidence of treatment-emergent adverse events as assessed by patient report.

SECONDARY OUTCOMES:
Change in Positive and Negative Symptom scale (PANSS) from Baseline to Day 14 | 14 days
  The PANSS is a 30-item clinician-rated instrument for assessing schizophrenia symptoms. It consists of 3 subscales: positive subscale (7 items), negative subscale (7 items), and general psychopathology subscale (16 items). For each item, symptom severity was rated on a 7-point scale, from 1=absent to 7=extreme. The PANSS total score for each participant was sum of the rating assigned to each of the 30 PANSS items, and ranged from 30 to 210 with a higher score indicating greater severity of symptoms. The reported measure is the change from baseline at until day 14.
Evaluate changes in NO bioavailability in breath from Baseline to Day 14 | 14 days
  Will measure change in NO bioavailability in breath using a Sievers NO Analyzer (NOA280i).
Change in blood levels of glutathione (GSH) from baseline to day 14. | 14 days
  Blood levels of glutathione (GSH) (uM) will be measured at baseline and day 14 via blood draw. Values of the this biomarker correspond to the bodies inflammatory and oxidative stress response. The results will be analyzed and compared from baseline to day 14 to measure for the effect of L-arginine and BH4 combination treatment on the body's inflammatory and oxidative stress response regulation.
Change in blood levels of high-sensitivity C reactive protein (hsCRP) from baseline to day 14. | 14 days
  Blood levels of high-sensitivity C reactive protein (hsCRP) (mg/L) will be measured at baseline and day 14 via blood draw. Values of the this biomarker correspond to the bodies inflammatory and oxidative stress response. The results will be analyzed and compared from baseline to day 14 to measure for the effect of L-arginine and BH4 combination treatment on the body's inflammatory and oxidative stress response regulation.
Change in blood levels of Tumor Necrosis Factor (TNF-α) from baseline to day 14. | 14 days
  Blood levels of Tumor Necrosis Factor (TNF-α) (pg/mL) will be measured at baseline and day 14 via blood draw. Values of the this biomarker correspond to the bodies inflammatory and oxidative stress response. The results will be analyzed and compared from baseline to day 14 to measure for the effect of L-arginine and BH4 combination treatment on the body's inflammatory and oxidative stress response regulation.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoduo Fan, Principal Investigator — UMass Medical School
Locations (1):
- UMass Medical School, Worcester, Massachusetts, United States